CLINICAL TRIAL: NCT05287724
Title: Pilot Studies Defining N-Acetyl Cysteine as a Treatment for Inhibiting Prurogenic Stimuli
Brief Title: Defining N-Acetyl Cysteine as a Treatment for Inhibiting Prurogenic Stimuli
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wright State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 07126
Record Dates: First submitted 2022-03-07; First posted 2022-03-18 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Pruritus; Skin Disorder
MeSH Terms: conditions — Pruritus; Skin Diseases | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- N-acetyl Cysteine then Placebo (Experimental): Subjects will be treated with N-acetyl cysteine twice daily for seven days. Subject will complete a minimum of 30-day washout period before crossing over to take the placebo.
  Interventions: Drug: N-acetyl cysteine; Drug: Placebo
- Placebo then N-acetyl Cysteine (Experimental): Subjects will be treated with placebo twice daily for seven days. Subject will complete a minimum of 30-day washout period before crossing over to take N-acetyl cysteine.
  Interventions: Drug: N-acetyl cysteine; Drug: Placebo

INTERVENTIONS:
Drug: N-acetyl cysteine — 1,500 mg twice daily for seven days
Drug: Placebo — Placebo taken twice daily for seven days

SUMMARY:
The objective of this double-blinded placebo-controlled cross-over study is to define the role of the over the counter agent, N-acetyl cysteine (NAC), in mitigating the development of pruritus (skin itching). The study is designed to have all subjects treated with a seven-day regimen of both NAC and placebo. NAC will be prescribed at a dose of 1,500 mg twice daily for seven days. Subjects will initially be randomly assigned (1:1) to either the NAC or placebo arm of the study, before crossing over to the opposite arm after completing a minimum of 30-day washout period. The study will encompass a period of approximately 11 weeks (about 2 and a half months).

ELIGIBILITY:
Inclusion Criteria:

* Males and Females
* All skin types (Fitzpatrick types I - VI)
* Age 18 - 40
* Able to comprehend procedures and risks

Exclusion Criteria:

* Currently taking immunosuppressive or immunomodulating or psychotropic medications.

This includes antihistamines and aspirin-like anti-inflammatory medications (NASIDs) for the past month.

* History of peripheral neuropathy, Charcot-Marie-Tooth, familial dysautonomia or heavy metal toxicity
* History of gastrointestinal abnormalities (including irritable bowel syndrome)
* History of inadequately controlled Diabetes Mellitus
* History of abnormal scarring
* History of skin infections within 6 weeks
* History of skin disease (atopic dermatitis, psoriasis, xerosis) or "sensitive skin"
* Pregnancy or nursing
* Other serious health issues, including liver or kidney disease

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-19 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Change in pain level from baseline with NAC. | 7 days
  The change will be assessed from the Skin Pain Visual Analogue Scale (0 = no skin pain to 10 = severe skin pain).
Change in pain level from baseline with placebo. | 7 days
  The change will be assessed from the Skin Pain Visual Analogue Scale (0 = no skin pain to 10 = severe skin pain).
Change in itch level from baseline with NAC. | 7 days
  The change will be assessed from the Skin Itch Visual Analogue Scale (0 = no skin itch to 10 = severe skin itch).
Change in itch level from baseline with placebo. | 7 days
  The change will be assessed from the Skin Itch Visual Analogue Scale (0 = no skin itch to 10 = severe skin itch).

CONTACTS AND LOCATIONS:
Overall Officials: Craig Rohan, MD, Principal Investigator — Wright State University
Locations (1):
- Wright State Physicians, Fairborn, Ohio, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/24/NCT05287724/ICF_000.pdf